CLINICAL TRIAL: NCT01555047
Title: Correlation Among Sperm DNA Fragmentation, Genitourinary Infection by Mycoplasma in Male and the Pregnancy Outcomes After IUI in Their Partner
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Feng Pan (Other)
Responsible Party: Sponsor-Investigator, Feng Pan, Clinical Attending Doctor, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NJU127
Record Dates: First submitted 2012-03-09; First posted 2012-03-15 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Mycoplasma
MeSH Terms: conditions — Mycoplasma Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- males who were not infected by mycoplasma (Active Comparator): 100 male patients whose spouse was going to conduct IUI, was not infected by mycoplasma.
  Interventions: Procedure: IUI
- infected by mycoplasma males (Experimental): 100 male patients whose spouse was going to conduct IUI, was infected by mycoplasma.
  Interventions: Procedure: IUI
- fertile males (No Intervention): 50 fertile males were chose as control samples

INTERVENTIONS:
Procedure: IUI — intrauterine insemination
  Arms: males who were not infected by mycoplasma
Procedure: IUI — intrauterine insemination
  Arms: infected by mycoplasma males

SUMMARY:
Genital ureaplasmas (Ureaplasma urealyticum and Ureaplasma parvum) and genital mycoplasmas (Mycoplasma hominis and Mycoplasma genitalium) are natural inhabitants of the male urethra contaminating the semen during ejaculation. However, these microorganisms, especially Ureaplasma urealyticum (Uu) and Mycoplasma hominis (Mh), are potentially pathogenic species playing an etiologic role in both genital infections and male infertility. Despite there are many consentaneous opinions about its relationship with infertility, its correlation with sperm regular parameters is still controversially. Sperm DNA damage can negatively influence fertilization rate, embryo cleavage rate, implantation rate, pregnancy and live birth rate, and is a novel indicator for intrauterine insemination (IUI) pregnancy rate and IVF or ICSI pregnancy loss rate. Until now, there were fewer clinical researches about the relationship among Uu and/or Mh infection, sperm DNA damage, and the IUI pregnancy rate. Thus, the investigators conduct this prospective study to investigate the relationship among them.

ELIGIBILITY:
Inclusion Criteria:

* Male with primary sterility with or without mycoplasma infection

Exclusion Criteria:

1. Combination with chlamydial infection
2. History of using hormone or cytotoxic drugs.
3. Having some other surgical diseases, such as genital tract infection or varicocele
4. Having some congenital diseases, such as Klinefelter and Y chromosome deficiency
5. Having some endocrine diseases, such as Kallmann, abnormality in pituitary gland, hyperthyroidism, hypercorticoidism, and so on
6. Patients' spouse had some diseases that could not carry out spontaneous pregnancy, such as tubal obstruction or ovulatory failure.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | up to 3 monthes after IUI

SECONDARY OUTCOMES:
sperm DNA fragmentation index (DFI) | one month before IUI